CLINICAL TRIAL: NCT03160833
Title: A Phase I/II, Open-label, Multi-center, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of HMPL-453 in Patients With Advanced Solid Malignancies
Brief Title: A Study of HMPL-453 in Patients With Advanced Solid Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-453-00CH1
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumor, Adult
Keywords: HMPL453; solid tumor; dose escalation

STUDY DESIGN:
Intervention Model Description: Open-label, Multi-center, Dose Escalation Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-453 (Experimental): Two strengths of HMPL-453 tablets (25 mg and 100 mg based on the free base) will be used for clinical studies. The drug products are coated tablets, which are packaged in white induction sealed HDPE (high-density polyethylene) bottles. HMPL-453 will be administered to patients as oral tablet(s) on a daily basis, until disease progression, intolerable toxicity, or death. Dose levels are to be potentially tested in this study include 50, 100, 200, 300, 400, and 500 mg/day
  Interventions: Drug: HMPL-453

INTERVENTIONS:
Drug: HMPL-453 — oral administrative

SUMMARY:
This is a dose escalation study consisting of two stages: Dose-escalation stage (stage 1): Patients will take a single dose of HMPL-453 on Day 1 and will be followed for one week for safety observations. After one week of observation, if no safety issues occur, patients can continue multiple dosing of HMPL-453 QD (quaque die) and start on the DLT (Dose Limited Toxicity) assessment cycles. Each cycle consists of 28-days. Patients are required to draw blood samples for PK and safety analysis at specific time points during the treatment; Dose-Expansion Stage (Stage 2): This stage is to further evaluate the safety, tolerability, PD (pharmacodynamics) profile, and preliminary anti-tumor activity of HMPL-453 at the RP2D (recommended phase 2 dose) in approximately 10 patients with advanced solid tumor.

DETAILED DESCRIPTION:
Dose-escalation stage (stage 1): Patients participating in the dose-escalation stage will take a single dose of HMPL-453 on Day 1 and will be followed for one week for safety observations. After one week of observation, if no safety issues occur, patients can continue multiple dosing of HMPL-453 QD and start on the DLT assessment cycles. Each cycle consists of 28-days. Patients are required to draw blood samples for PK and safety analysis at specific time points during the treatment.

The 3+3 design will be employed for the dose escalation and MTD ( maximum tolerated dose) determination. To limit the number of patients being exposed to potentially ineffective doses, one patient will be enrolled and dosed in the initial dose cohort. If there are no DLT or less than grade 2 toxicities of Common Terminology Criteria for Adverse Event ( CTC AE ) occur in the first treatment cycle, then the study will be escalated to the next dose cohort. Otherwise, the trial will revert to a standard 3+3 design.

Dose-Expansion Stage (Stage 2): This stage is to further evaluate the safety, tolerability, pharmacokinetics (PK) profile, and preliminary anti-tumor activity of HMPL-453 at the RP2D in approximately 60 patients with advanced solid tumor. Patients with FGFR ( Fibroblast Growth Factor Receptor) dysregulated advanced solid tumors, including but not limited to advanced urothelial bladder cancer, advanced cholangiocarcinoma (patients with cancers of the gallbladder or ampulla of Vater are not eligible) and others solid tumors are preferred to be enrolled.

Expansion stage will begin after dose-escalation stage is completed and the MTD/RP2D has been determined. Patients will receive HMPL-453 with 28-day treatment cycles until disease progression, death, intolerable toxicity, no longer benefiting from the study treatment per investigator's discretion, or withdrawal of consent, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* In the dose escalation stage, patients with locally advanced, or metastatic solid tumor who have failed, or intolerable to, standard therapies or for whom no standard therapies exist will be enrolled.
* In the dose expansion stage, patients with locally advanced, or metastatic solid tumor and FGFR dysregulation who have failed or intolerable to standard therapies or no standard therapies exist are to be enrolled.
* In the dose escalation stage: evaluable or measurable disease according to RECIST Version 1.1. In the dose expansion stage: measurable disease according to RECIST Version 1.1.
* Life expectancy of at least 12 weeks.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.

Exclusion Criteria:

* Prior or current treatment with any selective FGFR inhibitor.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs by the NCI CTCAE v4.03 | Cycle 1 (DLT assessment window 28 days)
  Incidence of DLTs by the NCI CTCAE v4.03

SECONDARY OUTCOMES:
Incidence of AEs and clinically significant laboratory abnormalities | From first dose to 30 days after last dose of study treatment
  incidence of any AEs associated to treatment
maximum plasma concentration (Cmax) | From first dose to day 56 of multiple dosing period
  maximum plasma concentration (Cmax) of HMP 453
time to reach maximum concentration (Tmax) | From first dose to day 56 of multiple dosing period
  time to reach maximum concentration (Tmax) of HMP 453
terminal half-life (t1/2) | From first dose to day 56 of multiple dosing period
  terminal half-life (t1/2) of HMP-453
area under the concentration-time curve (AUC0-t) | From first dose to day 56 of multiple dosing period
  area under the concentration-time curve (AUC0-t) of HMP453
apparent clearance (CL/F) | From first dose to day 56 of multiple dosing period
  apparent clearance (CL/F) of HMP 453
Serum phosphate level increases | From first dose to Day 21 of the last treatment cycle
  to evaluate the fluctuate level of Serum phosphate level
Objective response rate (ORR) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
  per RECIST
Duration of response (DoR) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
  from the date of response to progress or death
Disease Control Rate (DCR) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
  the response rate of PR (partial response) +CR(complete response) +SD （stable disease）
Change in tumor size | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
  per RECIST to evaluate the change of target and non-target lesions
Progression free survival (PFS) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
  Per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Weiss Yang, Doctor, Study Director — HMPL
Locations (2):
- China (2):
  - Beijing 307 Hospital, Beijing, Beijing Municipality
  - Cancer center of SYSU, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided